CLINICAL TRIAL: NCT05945875
Title: Official Title Targeted Dual Modality Imaging (TDMI) for Detection and Removal of Head and Neck Cancer
Brief Title: Evaluating the Use of Dual Imaging Techniques for Detection of Disease in Patients With Head and Neck Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Eben Rosenthal, Professor and Chair Department of Otolaryngology-, Vanderbilt-Ingram Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: VICC-EDHAN23204P; NCI-2023-05124 (Registry Identifier: NCI, Clinical Trials Reporting Program); 1R01CA266233-01A1 (NIH)
Record Dates: First submitted 2023-07-06; First posted 2023-07-14 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Head and Neck Squamous Cell Carcinoma; Recurrent Head and Neck Squamous Cell Carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Indium; Optical Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Diagnostic (panitumumab-IRDye800, 111In-panitumumab, SPECT/CT) (Experimental): Patients receive panitumumab-IRDye800 IV over 15 minutes followed by 111In-panitumumab IV on day 0. Patients then undergo SPECT/CT between days 1 and 5, prior to standard of care surgical resection with fluorescence imaging.
  Interventions: Drug: Panitumumab-IRDye800; Other: Indium In 111 Panitumumab; Procedure: Single Photon Emission Computed Tomography; Procedure: Computed Tomography; Procedure: Resection; Procedure: Fluorescence Imaging

INTERVENTIONS:
Drug: Panitumumab-IRDye800 — Given by IV
Other: Indium In 111 Panitumumab — Given by IV
Procedure: Single Photon Emission Computed Tomography — Undergo Single Photon Emission Computed Tomography
Procedure: Computed Tomography — Undergo Computed Tomography
Procedure: Resection — Undergo standard of care surgical resection
Procedure: Fluorescence Imaging — Undergo standard of care fluorescence imaging

SUMMARY:
This phase I trial evaluates the safety and effectiveness of using two imaging techniques, indium In 111 panitumumab (111In-panitumumab) with single photon emission computed tomography (SPECT)/computed tomography (CT) and panitumumab-IRDye800 fluorescence imaging during surgery (intraoperative), to detect disease in patients with head and neck cancer. 111In-panitumumab is an imaging agent made of a monoclonal antibody that has been labeled with a radioactive molecule called indium In 111. The agent targets and binds to receptors on tumor cells. This allows the cells to be visualized and assessed with SPECT/CT imaging techniques. SPECT is special type of CT scan in which a small amount of a radioactive drug is injected into a vein and a scanner is used to make detailed images of areas inside the body where the radioactive material is taken up by the cells. CT is an imaging technique for examining structures within the body by scanning them with x-rays and using a computer to construct a series of cross-sectional scans along a single axis. Panitumumab-IRDye800 is an imaging agent composed of panitumumab, a monoclonal antibody, linked to a fluorescent dye called IRDye800. Upon administration, panitumumab-IRDye800 targets and binds to receptors on tumor cells. This allows the tumor cells to be detected using fluorescence imaging during surgery. Adding 111In-panitumumab SPECT/CT imaging to intraoperative panitumumab-IRDye800 fluorescence imaging may be more effective at detecting disease in patients with head and neck cancer.

DETAILED DESCRIPTION:
Primary Objective:

- Assess the safety of the dual modality imaging (DMI) molecular agents, indium In 111 panitumumab (111In-panitumumab) and panitumumab-IRDye800, in patients with head and neck squamous cell carcinoma (HNSCC).

SECONDARY OBJECTIVES:

* Determine the sensitivity and specificity of 111In-panitumumab and panitumumab-IRDye800 for the detection of subclinical disease during primary tumor removal.
* Determine sensitivity and specificity of 111In-panitumumab and panitumumab-IRDye800 for detection of lymph nodes.

OUTLINE:

Patients receive panitumumab-IRDye800 intravenously (IV) over 15 minutes followed by 111In-panitumumab IV on day 0. Patients then undergo SPECT/CT between days 1 and 5, prior to standard of care surgical resection with fluorescence imaging.

After completion of study intervention, patients are followed up at day 15.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 19 years
* Biopsy-confirmed diagnosis of squamous cell carcinoma of the head and neck
* Subjects diagnosed with any T stage, any subsite within the head and neck that are scheduled to undergo surgical resection and neck dissection. Subjects with recurrent disease or a new primary will be allowed
* Planned standard of care elective neck dissection for a cN0 or node- positive disease. Clinical node- positive disease will be defined as metastasis in a single, ipsilateral lymph node, 3 cm or less in greatest dimension by clinical exam, cross sectional imaging or metabolic imaging
* Hemoglobin >= 9 gm/dL
* White blood cell count > 3000/mm^3
* Platelet count >= 100,000/mm^3
* Serum creatinine =< 1.5 times upper reference range
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Myocardial infarction (MI); cerebrovascular accident (CVA); uncontrolled congestive heart failure (CHF); significant liver disease; or unstable angina within 6 months prior to enrollment
* Evidence of QT prolongation on pretreatment electrocardiogram (ECG) (greater than 440 ms in males or greater than 450 ms in females)
* History of infusion reactions to monoclonal antibody therapies
* History of allergies to iodine
* Pregnant or breastfeeding
* Magnesium or potassium lower than the normal institutional values
* Subjects receiving class IA (quinidine, procainamide) or class III (dofetilide, amiodarone, sotalol) antiarrhythmic agents
* Subjects with a history or evidence of interstitial pneumonitis or pulmonary fibrosis
* Severe renal disease or anuria
* Thyroid stimulating hormone (TSH) > 13 micro international units/mL

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-10-03 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of grade 2 or higher adverse events | Up to day 15
  Will assess the number of grade 2 or higher adverse events determined to be significant and definitely or probably related to the study drugs. Adverse events will be evaluated using the Common Terminology Criteria for Adverse Events version 5.0 and summarized by grade, severity, and type.

SECONDARY OUTCOMES:
Sensitivity of 111In-panitumumab and panitumumab-IRDy800 for the detection of tumor-involved margins | Up to 4 years
  Detection of a positive margin defined as 1) presence of tumor within 5 mm of the cut surface of the specimen by using fluorescence imaging and 2) residual tumor present after removal of primary specimen by using fluorescence imaging and nuclear (gamma) signal in the wound bed. Findings will be compared to final histopathology as a reference standard. Presence of positive margin and residual tumor in the wound bed will be analyzed separately. Will calculate sensitivity with its 95% confidence interval. Will further perform McNemar's agreement test to examine whether there is any evidence of disagreement between these two sets of results.
Specificity of 111In-panitumumab and panitumumab-IRDy800 for the detection of tumor-involved margins | Up to 4 years
  Detection of a positive margin defined as 1) presence of tumor within 5 mm of the cut surface of the specimen by using fluorescence imaging and 2) residual tumor present after removal of primary specimen by using fluorescence imaging and nuclear (gamma) signal in the wound bed. Findings will be compared to final histopathology as a reference standard. Presence of positive margin and residual tumor in the wound bed will be analyzed separately. Will calculate specificity with its 95% confidence interval. Will further perform McNemar's agreement test to examine whether there is any evidence of disagreement between these two sets of results.
Sensitivity of 111In-panitumumab and panitumumab-IRDy800 for the detection of tumor-involved lymph nodes | Up to 4 years
  Intraoperatively, the number and location of tumor-positive lymph nodes will be determined using gamma signal and fluorescence imaging in the same format that surgeons have used during sentinel node mapping. Will perform near infrared fluorescence imaging and determine if these fluorescent lymph node(s) contain 111In-panitumumab via gamma tracing. All lymph nodes will be compared to gold standard histopathology for presence of disease.
Specificity of 111In-panitumumab and panitumumab-IRDy800 for the detection of tumor-involved lymph nodes | Up to 4 years
  Intraoperatively, the number and location of tumor-positive lymph nodes will be determined using gamma signal and fluorescence imaging in the same format that surgeons have used during sentinel node mapping. Will perform near infrared fluorescence imaging and determine if these fluorescent lymph node(s) contain 111In-panitumumab via gamma tracing. All lymph nodes will be compared to gold standard histopathology for presence of disease.

CONTACTS AND LOCATIONS:
Overall Officials: Eben Rosenthal, MD, Principal Investigator — Vanderbilt University/Ingram Cancer Center
Locations (1):
- Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Burns CR, Mattingly AS, Ely K, Radevic A, Meeks N, Zaidi SMA, Brown B, Vasiukov G, Topf M, Rosenthal E. Intraoperative Molecular Imaging Can Detect Large Nerve Perineural Invasion: A Case Report. Head Neck. 2026 Jan 7. doi: 10.1002/hed.70160. Online ahead of print. PMID 41498537

DOCUMENTS (1):
  • Informed Consent Form (2025-01-16): https://cdn.clinicaltrials.gov/large-docs/75/NCT05945875/ICF_000.pdf